CLINICAL TRIAL: NCT01419535
Title: Effects of the Glucocorticoid Antagonist, Mifepristone, on Glucose Intolerance in Obese and Overweight Individuals
Brief Title: Mifepristone Effects on Glucose Intolerance in Obese/Overweight Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 110208; 11-CH-0208 (Other: NIH); ZIADK075121 (NIH)
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Endocrine Disease; Diabetes
Keywords: Metabolism; Cortisol; Hypercortisolism; Glucose Intolerance
MeSH Terms: conditions — Endocrine System Diseases; Diabetes Mellitus; Cushing Syndrome; Glucose Intolerance | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Mifepristone, then Placebo (Experimental): Participants first received Mifepristone 50mg tablet every six hours for nine days. After a washout period of no fewer than 6 but no more than 8 weeks, they then received Placebo tablet (matching mifepristone 50 mg) every six hours for nine days.
  Interventions: Drug: Mifepristone; Drug: Placebo
- Placebo, then Mifepristone (Experimental): Participants first received Placebo tablet (matching mifepristone 50 mg) every six hours for nine days. After a washout period of no fewer than 6 but no more than 8 weeks, they then received Mifepristone 50 mg tablet every six hours for nine days.
  Interventions: Drug: Mifepristone; Drug: Placebo

INTERVENTIONS:
Drug: Mifepristone — Mifepristone 50mg tablet by mouth every six hours for nine days.
  Other Names: 55245; 11β-[p-(Dimethylamino)phenyl]-17α-(1-propynyl)estra-4,9-dien-17β-ol-3-one
Drug: Placebo — Placebo (matching mifepristone 50mg tablet) by mouth every six hours for nine days.
  Other Names: inert look-alike tablet

SUMMARY:
Background:

* Metabolic syndrome is a name given to a group of factors that tend to occur together. These risk factors include central obesity (extra weight around the middle of the body) and high blood pressure and blood sugar levels. They also include low levels of HDL ("good cholesterol") and high triglyceride levels. A person is said to have metabolic syndrome if they have three or more of the above risk factors. People with metabolic syndrome are at increased risk for type 2 diabetes, stroke, and heart disease.
* Cortisol, a hormone produced by the adrenal glands, is an important regulator of metabolism. People with central obesity and metabolic syndrome may have higher than normal cortisol levels that the body cannot regulate properly. Abnormal cortisol levels may play an important role in metabolic syndrome. Mifepristone is a drug that blocks cortisol. Researchers are interested in studying its effects on metabolic syndrome.

Objectives:

- To study the effects of short-term mifepristone treatment for metabolic syndrome.

Eligibility:

- Men and Women between 35 and 70 years of age are overweight or obese, and have abnormal glucose and triglyceride levels.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests.
* Participants will be admitted to the metabolic unit at the National Institutes of Health Clinical Center for the first 3 days of the study:
* Day 1: Body measurements (height, weight, waist, hip, and neck) and blood pressure tests. Also, 24 hours of regular blood draws and 24-hour urine collection to monitor regular daily cortisol levels.
* Day 2: Glucose/insulin infusion test to measure blood sugar levels.
* Day 3: Infusion of cortisol-like compounds and then regular blood draws for about 3 hours to evaluate how cortisol is metabolized.
* At the end of Day 3, participants will receive mifepristone or a look-alike capsule to take for 7 days at home.
* After 7 days, participants will return to the metabolic unit to repeat the Day 1 and Day 2 study procedures. They will continue to take mifepristone.
* One week after the second set of study tests, participants will return for a brief physical exam and blood tests.
* The study procedures will be repeated after 6 to 8 weeks, with the other study drug.

DETAILED DESCRIPTION:
The hormone cortisol is a key regulator of metabolism that influences the use of glucose (sugar) and fat as fuels. Persistently increased cortisol levels, as in Cushing s syndrome, lead to obesity, type 2 diabetes mellitus and lipid abnormalities including elevated triglyceride levels and low high-density lipoprotein (HDL) levels. These same disorders are also present in patients without Cushing s syndrome, suggesting that cortisol may be involved in their pathogenesis. Mifepristone is a cortisol-like drug that blocks cortisol action in the body. It can reverse lipid abnormalities, diabetes and obesity in Cushing s syndrome patients but its effects on these conditions have not been tested in patients without the syndrome.

The long-term aim of this clinical trial is to evaluate the ability of mifepristone to reverse or improve glucose intolerance, dyslipidemia, hypertension and weight gain. An initial 7-day prospective, randomized, placebo-controlled, crossover study is proposed here to look at the effect of short-term administration of oral mifepristone or placebo on glucose intolerance. Given that there are no human data available on the effect of mifepristone on insulin sensitivity, this will be a pilot study of 15 subjects. Data from this study will then be used to design a larger trial to evaluate long-term effects on blood pressure and weight, as well as glucose and triglyceride control.

Overweight or obese subjects with abnormal glucose tolerance will undergo each of the two treatments in a randomized order, including mifepristone by mouth and a look-alike inert tablet by mouth. Each treatment study will include two or three days of baseline tests that will be repeated after seven days of treatment. Treatments will be separated by at least six and no more than eight weeks. The tests will include blood drawing, urine collection, administration of glucose and insulin by vein, and a cortisol-like material to evaluate the metabolism of cortisol and a related hormone, corticosterone.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Men and women 35 - 70 years of age
  2. Subjects will be overweight or obese, with body mass index (BMI) ranging from 25 - 37 kg/m2.
  3. Subjects will have either impaired fasting glucose (greater than or equal to 100 mg/dL) or a 2-hour glucose value greater than or equal to 140 mg/dl during an oral glucose tolerance test (OGTT).

     OR

     Mild diabetes defined as patients with a Hemoglobin A1C (HbA1C) less than or equal to 7% on no medications (diet-controlled) or on a stable dose of metformin and no other hypoglycemic agents for greater than or equal to 3 months before study entry.
  4. Willing and able to comply with study requirements.

EXCLUSION CRITERIA:

1. Pregnancy and lactation
2. Diabetes requiring pharmacologic treatment. Diagnosis of diabetes will be based on the 2011 American Diabetes Association guidelines: HbA1C greater than or equal to 6.5%, fasting plasma glucose greater than or equal to 126 mg/dl, 2-hour glucose greater than or equal to 200 mg/dl during an OGTT, or a random blood glucose greater than or equal to 200 mg/dl along with classic symptoms of hyperglycemia (34)
3. Uncontrolled hypertension (blood pressure greater than or equal to 180/110 mmHg)
4. Current unstable medical conditions including clinically significant impaired cardiac function (Stage III and IV Cardiac failure), cardiac ischemia, severe respiratory insufficiency requiring oxygen therapy as assessed on history and/or physical exam
5. Liver function tests (alanine aminotransferase (ALT), aspartate aminotransferase (AST) more than 3-times the upper normal limit
6. Severe renal impairment (creatinine clearance < 30 ml/min)
7. Evidence of human immunodeficiency virus (HIV) based on history and physical examination and/or known positive HIV antibodies
8. Evidence of hepatitis C based on history and physical examination and/or known positive hepatitis C (HCV) antibody
9. History of hemorrhagic disorders or on anticoagulants
10. History of endometrial cancer, endometrial hyperplasia, unexplained vaginal bleeding, or endometrial thickness greater than 6 mm
11. Change in dose of lipid-lowering medications (including 3-hydroxy-3-methyl-glutaryl-coenzyme A reductase (HMG Co-A) inhibitors , fibrates, niacin, ezetimibe, and over-the-counter fish oil supplements) within one month of study entry and during the study period
12. Current administration of medications known to be strong CYP3A4 inhibitors including ketoconazole, itraconazole, and erythromycin
13. Use of herbal supplements or grapefruit juice within 14 days of study drug initiation
14. Use of medications or dietary supplements that inhibit or induce CYP3A4 activity within 14 days of study drug initiation
15. Use of oral, injectable, or inhaled glucocorticoids or megestrol in the past six months
16. Use of estrogen-containing hormone therapy
17. Potential pseudocushing's states: depression or intake of > 2 alcoholic drinks a day. Subjects will be screened for depression using the well-validated physician health questionnaire-9 (PHQ-9) with a score cut-off of greater than or equal to 10 for moderate depression (35).
18. Subjects who are actively dieting or are in a weight loss program
19. Midnight salivary cortisol > 100 ng/dl on two separate occasions
20. Untreated thyroid dysfunction (thyroid stimulating hormone and Free thyroxine (FT4) not within normal range). If abnormal on screening labs, they will be repeated to confirm that not due to lab error or non-thyroidal illness.
21. Moderate to severe anemia (hemoglobin < 10 g/dl)
22. Blood donation of more than 500 ml within one month prior to study enrollment
23. Subjects with a prolonged corrected Q-T interval (QTc) on electrocardiogram
24. Unable to give informed consent

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-11-29 (Actual); Primary Completion 2015-11-24 (Actual); Study Completion 2015-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, individual participant data will be shared with other investigators
Supporting Information: CSR
Time Frame: Upon publication, for two years
Access Criteria: plan for data use

REFERENCES:
- [Background] Pivonello R, Faggiano A, Lombardi G, Colao A. The metabolic syndrome and cardiovascular risk in Cushing's syndrome. Endocrinol Metab Clin North Am. 2005 Jun;34(2):327-39, viii. doi: 10.1016/j.ecl.2005.01.010. PMID 15850845
- [Background] Anagnostis P, Athyros VG, Tziomalos K, Karagiannis A, Mikhailidis DP. Clinical review: The pathogenetic role of cortisol in the metabolic syndrome: a hypothesis. J Clin Endocrinol Metab. 2009 Aug;94(8):2692-701. doi: 10.1210/jc.2009-0370. Epub 2009 May 26. PMID 19470627
- [Background] Pasquali R, Vicennati V, Cacciari M, Pagotto U. The hypothalamic-pituitary-adrenal axis activity in obesity and the metabolic syndrome. Ann N Y Acad Sci. 2006 Nov;1083:111-28. doi: 10.1196/annals.1367.009. PMID 17148736
- [Derived] Gubbi S, Muniyappa R, Sharma ST, Grewal S, McGlotten R, Nieman LK. Mifepristone Improves Adipose Tissue Insulin Sensitivity in Insulin Resistant Individuals. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1501-1515. doi: 10.1210/clinem/dgab046. PMID 33507248
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-CH-0208.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited to the study by advertisements and fliers. Sixty-three adults were evaluated at the single study site (the NIH Clinical Center) after providing informed consent. The first subject consented on November 11, 2011 and the final subject consented on April 16, 2015.
Pre-assignment Details: Forty-four subjects were excluded; 31 had a normal oral glucose tolerance test and fasting glucose level, 2 exceeded BMI criterion, 2 exceeded HbA1C criterion, 2 had depression, and seven subjects had one of the following exclusion criteria: required insulin, <35 years old, memory problems/compliance, abnormal thyroid function, drop out after screening, abnormal late night salivary cortisol, failure to complete screening. The remaining 19 subjects were randomized.
Period: Overall Study
Arm/Group | Mifepristone, Then Placebo | Placebo, Then Mifepristone
Started | 9 | 10
Completed | 8 | 8
Not Completed | 1 | 2
Not completed — could not maintain iv line | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone, Then Placebo | Placebo, Then Mifepristone | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (6.5) | 52.8 (8.9) | 54.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Weight [Mean (Standard Deviation); unit: kg] | 92.8 (15.8) | 102 (15.9) | 97.2 (16.0)
Body mass index [Mean (Standard Deviation); unit: kg/M^2] | 30.8 (4.12) | 34.0 (2.37) | 32.4 (4.12)
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 124 (16.1) | 133 (10.5) | 128 (13.9)
diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 77.6 (4.7) | 76.9 (9.9) | 77.3 (7.5)
total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 177.9 (59.0) | 184.3 (53.8) | 181.1 (54.6)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 51.1 (7.5) | 40.0 (8.6) | 45.6 (9.7)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 104.9 (41.3) | 108.3 (41.0) | 106.6 (40.1)
triglycerides [Mean (Standard Deviation); unit: mg/dL] | 108.8 (88.3) | 180.0 (92.3) | 144.4 (94.7)
free fatty acids [Mean (Standard Deviation); unit: mg/dL] | 0.62 (0.18) | 0.54 (0.23) | 0.60 (0.19)
fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 101.0 (5.8) | 108.1 (20.6) | 104.6 (15.0)
fasting insulin [Mean (Standard Deviation); unit: pmol/L] | 75.7 (35.4) | 143.1 (43.3) | 109 (51.8)
A1C [Mean (Standard Deviation); unit: percent] | 5.9 (0.35) | 6.3 (0.49) | 6.1 (0.45)
Urine free cortisol [Mean (Standard Deviation); unit: ug/dl] | 27.8 (23.0) | 18.1 (7.2) | 22.9 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity Index
Description: insulin sensitivity index based on the effect of insulin on glucose during frequently sampled intravenous glucose tolerance test (FSIVGTT)
Time Frame: Nine days
Population: 2 subjects in each group missing data due to iv line problems
Measure: Mean (Standard Deviation); unit: min-1·μU·ml-1
Groups:
- Post-mifepristone: All subjects tested after mifepristone administration, compared to baseline
- Post-placebo: all subjects tested after placebo administration, compared to baseline
Arm/Group | Post-mifepristone | Post-placebo
Number analyzed (Participants) | 16 | 16
min-1·μU·ml-1 | 1.49 (1.17) | 1.41 (0.87)
Statistical Analysis 1: Comparison: Post-mifepristone vs Post-placebo; Test type: Superiority; p = 0.60, ANOVA; Repeated measures were analyzed by repeated-measures ANOVA including treatment group, time, and treatment*time interaction as factors

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: fasting plasma glucose after study agent compared to baseline
Time Frame: Nine days
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Post-mifepristone | Post-placebo
Number analyzed (Participants) | 16 | 16
mg/dL | 100.4 (5.3) | 107.8 (15.7)
Statistical Analysis 1: Comparison: Post-mifepristone vs Post-placebo; Test type: Superiority; p < 0.001, ANOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Fasting Insulin Levels
Description: Fasting insulin after study agent administration compared to baseline
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Post-mifepristone | Post-placebo
Number analyzed (Participants) | 16 | 16
pmol/L | 95.6 (76.1) | 142.8 (102.2)
Statistical Analysis 1: Comparison: Post-mifepristone vs Post-placebo; Test type: Superiority; p < 0.001, ANOVA; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR is an index of insulin resistance, measured as glucose in mmol/L x insulin in mIU/mL)/22.5. HOMA-IR > 2.5 indicates insulin resistance.
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post-mifepristone | Post-placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 3.58 (3.27) | 5.78 (4.92)
Statistical Analysis 1: Comparison: Post-mifepristone vs Post-placebo; Test type: Superiority; p < 0.001, ANOVA; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Adipose-tissue Insulin Resistance Index (Adipo-IR)
Description: The adipose tissue insulin resistance index (Adipo-IR), a surrogate measure for fasting adipose-tissue insulin resistance, was calculated as the product of fasting insulin and fasting free fatty acids (FFA)
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: mmol/l·μU/l
Arm/Group | Post-mifepristone | Post-placebo
Number analyzed (Participants) | 16 | 16
mmol/l·μU/l | 49.9 (45.9) | 65.5 (43.8)
Statistical Analysis 1: Comparison: Post-mifepristone vs Post-placebo; Test type: Superiority; p = 0.004, ANOVA; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Adipose-tissue Insulin Sensitivity Index (Adipo-SI)
Description: The Adipo-SI was calculated as ratio of the slope of the linear decrease in natural log transformed FFA [Ln (FFA) slope] during the first 90 minutes of the FSIVGTT and the area under the curve (AUC) of insulin during that 90-minute period (AUC Insulin 0-90 min).
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: ln(mmol /uU/mL*min)*10^8
Arm/Group | Post-mifepristone | Post-placebo
Number analyzed (Participants) | 16 | 16
ln(mmol /uU/mL*min)*10^8 | 61.7 (32.9) | 42.8 (23.9)
Statistical Analysis 1: Comparison: Post-mifepristone vs Post-placebo; Test type: Superiority; p = 0.002, ANOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Subjects returned for safety labs and discussion of any adverse events on approximately day 19 and day 33 after discontinuation of study agents.
Arm/Group | Post-mifepristone | Post-placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-mifepristone (N=16) | Post-placebo (N=16)
abnormal blood chemistry (Hepatobiliary disorders) | 0 (0) | 2 (2) — elevated alanine transferase less than one-fold above the upper limit of normal, resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT01419535/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT01419535/ICF_001.pdf